CLINICAL TRIAL: NCT06285669
Title: Effects of Kinesio Taping Applications on Diaphragm, Respiratory Muscles and Chest Wall In Very Preterm Infants On Non-invasive Ventilation
Brief Title: Effects of Kinesiotaping on Respiratory Muscles in Very Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Associate Proffessor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA18/35
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Preterm; Premature; Infant, Newborn, Diseases; Respiratory Distress Syndrome; Neonatal Respiratory Distress
Keywords: respiratory distress syndrome; preterm infant; kinesiotaping; pulmonary function
MeSH Terms: conditions — Premature Birth; Infant, Newborn, Diseases; Respiratory Distress Syndrome; Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Kinesio-Taping Application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotape (Experimental): Kinesio taping was applied by a single physiotherapist to support the intercostal muscles,and, the diaphragm and facilitatory method was used on the respiratory muscles
  Interventions: Other: kinesiotaping application
- Control (No Intervention): This group didn't take kinesiotape application

INTERVENTIONS:
Other: kinesiotaping application — kinesiotaping application
  Arms: kinesiotape

SUMMARY:
This study aimed to evaluate the effects of kinesio taping on blood gas parameters, respiratory rate, heart rate, oxygen saturation, and pressure limits in preterm infants with RDS who are on NIV. It is hypothesized that the application of kinesio taping to the chest area of preterm infants may improve respiratory functions and oxygenation at the alveolar level, leading to decreased work of breathing, reduced respiratory rate, and improved neonatal stability by promoting respiratory mechanics and enhancing chest expansion.

DETAILED DESCRIPTION:
Very preterm infants are at high risk of respiratory distress syndrome (RDS), due to surfactant deficiency and weak respiratory muscles. This condition can contribute to respiratory workload and irregular breathing. This study aimed to investigate the effects of Kinesio kinesio-taping technique on the respiratory muscles and diaphragm in very preterm infants undergoing non-invasive.

Twenty-six preterm infants born before the 32nd gestational week and requiring non-invasive ventilation (NIV) support due to RDS, were randomly divided into 2 groups as Kinesio taping group and control group. Kinesio taping was applied by a single physiotherapist to support the intercostal muscles,and, the diaphragm and facilitatory method was used on the respiratory muscles. Kinesio taping was removed just after preterm infants were weaned from noninvasive ventilation. Blood gas parameters, respiratory rate, heart rate, FiO2, FiO2/pO2 ratio, PIP, PEEP values, and length of stay in NIV were recorded before and after 3 days of KT application.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants diagnosed with RDS
* Preterm Infants born under 32 weeks of gestation

Exclusion Criteria:

* Sepsis,
* necrotizing enterocolitis,
* metabolic disease,
* severe congenital malformations of the chest and abdominal walls,
* congenital heart disease,
* major congenital anomalies

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Level of pH | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Comuk Balci, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Nilay Çömük Balci, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No